CLINICAL TRIAL: NCT00943709
Title: Effects of Intensive Glycemic Control on Infectious Morbidity In Patients With Acute Leukemia
Brief Title: Intensive Glycemic Control on Infectious Morbidity In Patients With Acute Leukemia
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: lack of accrual
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Sanofi (Industry)
Responsible Party: Sponsor
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 060601; AVENTIS-CINJ-060601; 0220070268 (Other: IRB Number); CDR0000648982; P30CA072720 (NIH)
Record Dates: First submitted 2009-07-21; First posted 2009-07-22 (Estimated); Last update posted 2013-08-30 (Estimated); Status verified 2013-08

CONDITIONS: Hyperglycemia; Leukemia
Keywords: hyperglycemia; recurrent adult acute lymphoblastic leukemia; untreated adult acute lymphoblastic leukemia; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); recurrent adult acute myeloid leukemia; untreated adult acute myeloid leukemia
MeSH Terms: conditions — Hyperglycemia; Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Congenital Abnormalities; Leukemia, Myeloid, Acute | interventions — Insulin Glargine; Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Patients with goal blood glucose 80-14 mg/dL receive the Robert Wood Johnson Hospital IV insulin infusion protocol followed by insulin glargine and insulin glulisine (Apidra™) subcutaneously for 4 weeks.
  Interventions: Biological: insulin glargine recombinant; Drug: therapeutic insulin
- Arm II (Active Comparator): Patients with goal blood glucose < 250 mg/dL are started on subcutaneous insulin sliding scale at the discretion of the treating physician with blood glucose monitoring and adjustment according to the insulin sliding scale.
  Interventions: Biological: insulin glargine recombinant; Drug: therapeutic insulin

INTERVENTIONS:
Biological: insulin glargine recombinant — Given subcutaneously
Drug: therapeutic insulin — Given subcutaneously

SUMMARY:
RATIONALE: Controlling blood sugar levels may be effective in preventing infections in patients receiving chemotherapy for acute myeloid leukemia or acute lymphoblastic leukemia.

PURPOSE: This randomized phase I trial is studying how well controlling blood sugar levels works in preventing infection in patients with acute myeloid leukemia or acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine whether intensive glycemic control over an eight week time period will decrease the incidence of infections from initiation of chemotherapy treatment in patients with acute myeloid leukemia or acute lymphoblastic leukemia.

Secondary

* To compare the number of episodes of infection.
* To compare the duration of neutropenia.
* To compare the number of days of bacteremia/fungemia.
* To compare the number of days of fever.
* To compare the duration of nutrition.
* To compare the duration of mucositis.
* To compare the duration of hospital stay.
* To compare the duration of antibiotic use.
* To compare the incidence of thromboembolic events.
* To compare body weight changes.
* To compare the median survival.
* To compare the remission rate with induction or salvage chemotherapy.
* To conduct comparative analysis between intervention and standard of care groups of mean daily capillary blood glucose monitoring.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

* Arm I (intensive glycemic control): Patients with goal blood glucose 80-140 mg/dL receive the Robert Wood Johnson University Hospital IV insulin infusion protocol to maintain blood glucoses in the target range. Beginning 24 hours after maintenance of oral or enteral feedings patients receive an intensive regimen of insulin glargine and insulin glulisine (Apidra™) subcutaneously for 4 weeks as needed. Patients may also receive insulin in the total parenteral nutrition (TPN) mixture.
* Arm II (standard care control): Patients with goal blood glucose < 250 mg/dL are started on subcutaneous insulin sliding scale at the discretion of the treating physician with blood glucose monitoring and adjustment according to the insulin sliding scale. Insulin may also be added to TPN if needed at the investigator's discretion.

After completion of study treatment, patients are followed up for 4 weeks.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed acute myeloid leukemia or acute lymphoid leukemia

  * Newly diagnosed or relapsed disease
* Undergoing induction or salvage chemotherapy treatment
* Must demonstrate 2 random blood sugars of ≥ 140 mg/dL while on total parenteral nutrition (TPN) OR 2 preprandial sugars of ≥ 140 mg/dL if patient is not on TPN

PATIENT CHARACTERISTICS:

* ECOG performance status 0-3
* Not pregnant or nursing
* Negative pregnancy test
* Prior diagnosis of diabetes mellitus allowed
* No known history of an allergy to insulin
* No documented active infection

PRIOR CONCURRENT THERAPY:

* Concurrent corticosteroids allowed
* No concurrent oral hypoglycemic agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-05; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Incidence of new infections | 4 years

SECONDARY OUTCOMES:
Number of episodes of infection | 4 years
Duration of neutropenia | 4 years
Number of days of bacteremia/fungemia | 4 years
Number of days of fever | 4 years
Duration of nutrition | 4 years
Duration of mucositis | 4 years
Duration of hospital stay | 4 years
Duration of antibiotic use | 4 years
Incidence of thromboembolic events | 4 years
Body weight changes | 4 years
Median survival | 4 years
Remission rate with induction or salvage chemotherapy | 4 years
Comparative analysis between intervention and standard of care groups of mean daily capillary blood glucose monitoring | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Mecide Gharibo, MD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (1):
- Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey, United States